CLINICAL TRIAL: NCT00359723
Title: Subacute Trial of Methylphenidate in Parkinson's Disease
Brief Title: Methylphenidate and Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, John G. Nutt, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00000959; R01NS021062 (NIH)
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; methylphenidate; Ritalin; MPD
MeSH Terms: conditions — Parkinson Disease | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Methylphenidate 0.4 mg/kg TID followed by placebo TID (Experimental): As above
  Interventions: Drug: methylphenidate
- Placebo TID followed by methylphenidate 0.4 mg/kg TID (Experimental): As above
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: methylphenidate

SUMMARY:
The purpose of this trial is to determine if methylphenidate (MPD), a drug marketed in the U.S. to treat hyperactivity and narcolepsy, added to levodopa, will increase the beneficial effects of levodopa without bothersome side effects in people with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common disorder caused by the loss of dopamine-producing brain cells. The disorder is generally treated with levodopa combined with carbidopa. Nerve cells use levodopa to make dopamine. Carbidopa delays the conversion of levodopa into dopamine until it reaches the brain. Motor fluctuations (the wearing off effects of levodopa characterized by sometimes rapid changes between uncontrolled and normal movements) are a common, and often difficult to manage, source of disability in people with PD.

In this trial researchers will study the effects of methylphenidate (MPD), also known as Ritalin-a drug marketed in the U.S. to treat hyperactivity and narcolepsy-on carbidopa/levodopa and other antiparkinson medications taken orally by individuals with Parkinson's disease who experience motor fluctuations when they take levodopa. The overall goal of this project is to develop better symptomatic therapies for PD.

After 2 screening visits to the treatment clinic to evaluate the wearing "on" and "off" effects of levodopa, eligible participants will be scheduled for 3 admissions to the General Clinical Research Center at Oregon Health & Science University during which they randomly will receive the study drug, MPD, or placebo, along with their usual carbidopa/levodopa therapy and/or other antiparkinson medications. Also, participants will have their parkinsonism (tremor, rigidity, postural instability, and bradykinesia) rated and blood pressure and pulse measured at regular intervals.

Duration of the study for participants is about 3 weeks and includes 2 outpatient clinic visits (for screening) and 3 inpatient clinic visits (with overnight stays).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD treated with levodopa and experiencing motor fluctuations
* At least 21 years of age
* Male or female.

Exclusion Criteria:

* Cardiovascular disease, psychosis, extreme anxiety, dementia and other unstable medical conditions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-07; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Time "on" defined by tapping speed

CONTACTS AND LOCATIONS:
Overall Officials: John G. Nutt, MD, Principal Investigator — Professor of Neurology, Oregon Health Science University; Julie H. Carter, ANP, Principal Investigator — Oregon Health and Science University; Nichole T. Carlson, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Department of Neurology, OP-2, Oregon Health & Science University, 3181 SW Sam Jackson Park Road, Portland, Oregon, United States

REFERENCES:
- [Result] Nutt JG, Carter JH, Carlson NE. Effects of methylphenidate on response to oral levodopa: a double-blind clinical trial. Arch Neurol. 2007 Mar;64(3):319-23. doi: 10.1001/archneur.64.3.319. PMID 17353373